CLINICAL TRIAL: NCT03120221
Title: Iodine Status in Pregnant Women in Israel
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clalit Health Services (Other)
Responsible Party: Principal Investigator, Dr. Viviana Ostrovsky, Principal Investigator, Senior Physician, Endocrinology Department, Clalit Health Services
Other Study IDs: 0092-16-COM2
Record Dates: First submitted 2017-04-01; First posted 2017-04-19 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Iodine-Deficiency; Hypothyroidism
Keywords: Pregnancy; Iodine deficiency; Thyroid
MeSH Terms: conditions — Hypothyroidism; Thyroid Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- First trimester pregnant women
  Interventions: Diagnostic Test: Urine sample for iodine measurement

INTERVENTIONS:
Diagnostic Test: Urine sample for iodine measurement — Women will be required to give a urine sample for iodine measurement

SUMMARY:
Worldwide Data suggest that Iodine deficiency is a concern among healthy pregnant women. Thus, screening first trimester healthy pregnant women for iodine status is of clinical value for mother and child as iodine deficiency might have implications on thyroid function as well as pregnancy outcomes

DETAILED DESCRIPTION:
New emerging data suggest pregnant women in Israel are iodine deficient in the first trimester of pregnancy. This is of major concern as first trimester iodine sufficiency is critical for the development of the fetal brain. Our aim is to evaluate iodine consumption in first trimester pregnant women in Israel through dietary questioners, Urinary iodine samples and thyroid functions test assessed through blood samples. All data will be analyzed in a central lab.

ELIGIBILITY:
Inclusion Criteria: First trimester pregnant women with a singleton pregnancy

Exclusion Criteria:

1. Women with a known thyroid disease treated or untreated
2. Women who received contrast material in the year previous to the study
3. women with any chronic disease
4. Women who receive chronic medication not including vitamins

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Study Population: First trimester pregnant women in Israel
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2017-07-04 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of average iodine consumption in food | 1 year
  Iodine consumption will be evaluated trough detailed food questionnaires. Data will be quantified and reported in micrograms per day
Evaluation of urinary iodine concentration | 1 year
  Women will give a spot urine sample for urinary iodine concentration measurement. All data will be analyzed and reported in micrograms/L. Data obtained will be compared to World Health Organization requirements
Thyroid function test measurement | 1 year
  Thyroid function will be evaluated through blood tests in the first trimester of pregnancy. Data will be analyzed in accordance with local guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Viviana Ostrovsky, MD, Principal Investigator — Clalit Health Services
Locations (2):
- Israel (2):
  - Women Health Service, Ashdod
  - Women Health Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No